CLINICAL TRIAL: NCT02626195
Title: Prospective Study of Preoperative Nutritional Support in Malnutritional Pancreatobiliary Cancer Patients
Brief Title: Preoperative Nutritional Support in Malnutritional Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Sang-Jae Park, Head of Center for Liver Cancer, Chief of the Liver and Pancreatobiliary Cancer Branch, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-13-676
Record Dates: First submitted 2015-06-08; First posted 2015-12-10 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Cancer; Biliary Cancer; Malnutrition
Keywords: malnutrition; nutrition; nutritional support; hepatobiliary pancreatic cancer; hepatobiliary pancreatic surgery
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutritional support program apply (Experimental): Preoperative nutritional support program is given for 5 or more days preoperatively by nutritional support program.
  Interventions: Dietary Supplement: nutritional support program
- historical control group (No Intervention): Historical control group is that did not receiving

INTERVENTIONS:
Dietary Supplement: nutritional support program — Nutritional support program is briefly described below.
  Interval: 5-10 days Contents: admission is required
  * Calories: 30-35Kg, via enteral or parenteral
  * Protein: 1.2-1.5g/Kg
  * Lipid : 1-1.5g/Kg
  * Mineral and vitamins supply
  * Blood glucose control
  * Daily monitoring by dietician and specialized nurse
  Arms: nutritional support program apply

SUMMARY:
Malnutrition patients are known to have more postoperative complications and mortality. And most of hepatobiliary-pancreatic cancer surgeries accompany high postoperative morbidity and mortality rate. Therefore for the malnourished patients anticipating major surgery, preoperative nutritional support is recommended according to the ASPEN (American society of parenteral and enteral nutrition) and ESPEN (European society of parenteral and enteral nutrition) guideline. However there is no prospective trial to prove the clinical impact of preoperative nutritional support for malnourished patients.

The purpose of this study is to evaluate the clinical impact of preoperative nutritional support for malnourished cancer patients anticipating HBP surgery. Primary objective is to compare the complication rate and secondary object is to compare the quality of life, hospital stay and cost.

DETAILED DESCRIPTION:
This is single arm study with historical comparison. The historical control group did not receiving nutritional support. In previous results show that about 25% complication rates. Complication rates are expected in the group receiving nutritional support is less than 10 % ( previous studies (NCCNCS-11-460)).

For support group, preoperative nutritional support is given for 5 or more days preoperatively by nutritional support program. Nutritional support program is briefly described below.

Interval: 5-10 days Contents: admission is required

* Calories: 30-35Kg, via enteral or parenteral
* Protein: 1.2-1.5g/Kg
* Lipid : 1-1.5g/Kg
* Mineral and vitamins supply
* Blood glucose control
* Daily monitoring by dietician and specialized nurse

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in anticipating major surgery of hepatobiliary pancreatic cancer
2. Patients diagnosed with malnutrition (at least more than one)

   1. PG-SGA B or C
   2. Weight loss >10% within 6 month
   3. BMI <18.5
   4. Serum Albumin <3.0
3. Age less than 80 years old over 20 years old
4. Performance status (ECOG scale): 0-1
5. Adequate organ functions

   1. Hb ≥7.0 g/dl
   2. ANC ≥1,500/mm3
   3. PLT ≥80,000/mm3
   4. Liver function: AST/ALT ≤5×upper limit of normal
   5. Creatinine ≤2.0 ULN

Exclusion Criteria:

1. Biopsy, drainage tube insertion, and other minor surgery
2. palliative surgery
3. Serious illness or medical conditions, as follows;

   1. congestive heart failure (NYHA class III or IV)
   2. unstable angina or myocardial infarction within the past 6 months,
   3. significant arrhythmias requiring medication and conduction abnormality such as over 2nd degree AV block
   4. uncontrolled hypertension
   5. hepatic cirrhosis( ≥ Child class B)
   6. interstitial pneumonia, pulmonary adenomatosis
   7. psychiatric disorder that may interfere with and/or protocol compliance
   8. unstable diabetes mellitus
   9. uncontrolled ascites or pleural effusion
   10. active infection
4. Pregnancy
5. Any patients judged by the investigator to be unfit to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11-27 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
postoperative complication | at discharge. (expected the duration of hospital stay of postoperation is 4~6 weeks.)
  expected the duration of hospital stay of postoperation is 4~6 weeks.

SECONDARY OUTCOMES:
postoperative hospital stay | expected the duration of hospital stay of postoperation is 4~6 weeks.
  expected the duration of hospital stay of postoperation is 4~6 weeks.
quality of life | preoperative, postoperative 14days
  preoperative, postoperative 14days
postoperative cost( + nutritional support cost) | at discharge. (expected the duration of hospital stay of postoperation is 4~6 weeks.)
  expected the duration of hospital stay of postoperation is 4~6 weeks.

OTHER OUTCOMES:
immunologic change(CD4/CD8) after nutritional support | preoperative, postoperative 14days
  CD4/CD8, immunoglobulin G, M, A

CONTACTS AND LOCATIONS:
Overall Officials: SangJae Park, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No